CLINICAL TRIAL: NCT03009812
Title: Transverse Versus Longitudinal Uterine Incision in Abdominal Myomectomy
Brief Title: Transverse vs Longitudinal Incision in Myomectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, maii medhat nawara, Principle investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MY-789
Record Dates: First submitted 2017-01-01; First posted 2017-01-04 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Myoma;Uterus
MeSH Terms: conditions — Myofibroma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): 26 subjects who are planned for transverse uterine incision
  Interventions: Procedure: Transverse uterine incision
- Group 2 (Active Comparator): 26 subjects who are planned for longitudinal uterine incision
  Interventions: Procedure: Longitudinal uterine incision

INTERVENTIONS:
Procedure: Longitudinal uterine incision
  Arms: Group 2
Procedure: Transverse uterine incision
  Arms: Group 1

SUMMARY:
The Aim of the study is to compare between transverse and longitudinal uterine incision in abdominal myomectomy regarding intraoperative blood loss.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria for myomectomy as; abnormal uterine, pressure related symptoms, infertility and recurrent pregnancy loss in patients between 18 and 45 years old
2. Single myoma.
3. Women with BMI between 18.5-29.9 kg/m2.

Exclusion Criteria:

1. Pregnancy.
2. Patients with bleeding tendency
3. Previous laparotomies.
4. Patients with concomitant pelvic pathologies, such as ovarian cysts.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01-23 (Actual)

PRIMARY OUTCOMES:
Intraoperative blood loss | 1 year

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elguindy A, Hemeda H, Shawky ME, Elsenity M, Elsayed MA, Fahim A, Afifi K, Nawara M. Blood loss from transverse versus longitudinal uterine incision in abdominal myomectomy: a randomized controlled trial. BMC Womens Health. 2020 Dec 28;20(1):259. doi: 10.1186/s12905-020-01113-3. PMID 33357218